CLINICAL TRIAL: NCT02090517
Title: Evaluation of Laser Therapy Vs Electrosurgery For Nasal Telangiectasias Using A Novel Vascular Imaging Device
Brief Title: Laser Therapy Versus Electrosurgery For Nasal Telangiectasias
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was withdrawn because the university wanted to bill study patients for use of the laser.
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 430519; 430519 (Other: University of California, Davis)
Record Dates: First submitted 2013-12-04; First posted 2014-03-18 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Telangiectasis
Keywords: Nasal telangiectasis
MeSH Terms: conditions — Telangiectasis | interventions — Lasers, Dye

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Pulsed Dye Laser (Active Comparator): Subjects with multiple nose telangiectasias will be enrolled. One nose telangiectasia (of 5) will be treated with pulsed dye laser.
  Interventions: Device: Pulsed Dye Laser
- Long Pulsed Alexandrite Laser (Active Comparator): Subjects with multiple nose telangiectasias will be enrolled. One nose telangiectasia (of 5) will be treated with long pulsed alexandrite laser.
  Interventions: Device: Long Pulsed Alexandrite Laser
- Pulsed Dye Laser Plus Nd:YAG Laser (Active Comparator): Subjects with multiple nose telangiectasias will be enrolled. One nose telangiectasia (of 5) will be treated with pulsed dye laser plus Nd:YAG laser.
  Interventions: Device: Pulsed Dye Laser Plus Nd:YAG Laser
- Electrodesiccation (Active Comparator): Subjects with multiple nose telangiectasias will be enrolled. One nose telangiectasia (of 5) will be treated with electrodesiccation.
  Interventions: Procedure: Electrodesiccation
- No Treatment (No Intervention): Subjects with multiple nose telangiectasias will be enrolled. One nose telangiectasia (of 5) will receive no treatment.

INTERVENTIONS:
Device: Pulsed Dye Laser — Pulsed dye laser treatments will be performed with a 595 nanometer wavelength, 20 millisecond pulse duration, at 10 Joules/cm2, with a 10 millimeter spot size.
  Other Names: Pulsed dye laser treatments will be performed with a 595 nanometer wavelength, 20 millisecond pulse duration, at 10 Joules/cm2, with a 10 millimeter spot size.
  Arms: Pulsed Dye Laser
Device: Long Pulsed Alexandrite Laser — Alexandrite laser will be used with a 755 nanometer wavelength, 40 millisecond pulse duration, at 88Joules/cm2, with a 6 millimeter spot size.
  Arms: Long Pulsed Alexandrite Laser
Device: Pulsed Dye Laser Plus Nd:YAG Laser — The Cynergy with MultiPlex will be used with a multiplex mode system with a pulse dye laser at 585 nanometer wavelength, 20 milliseconds pulse duration, at 7 Joules/cm2 with a 7 millimeter spot size, with a short delay, followed by a Nd:YAG 1064 nanometer wavelength, 20 millisecond pulse duration, at 50 Joules/cm2 with a 7 millimeter spot size.
  Arms: Pulsed Dye Laser Plus Nd:YAG Laser
Procedure: Electrodesiccation — A curette is used to scrape off the cancer down to the dermis. The scraping is then paused while an electrosurgical device like a hyfrecator is used next. Electrodesiccation is performed over the raw surgical ulcer to denature a layer of the dermis and the curette is used again over the surgical ulcer to remove denatured dermis down to living tissue.
  Arms: Electrodesiccation

SUMMARY:
The aim of this study is to compare the efficacy of various treatment options for eliminating nasal telangiectasias. The study will compare the outcome of treating nasal telangiectasias with the following; no treatment (control site), alexandrite laser, pulsed dye laser, combination pulsed dye laser and Nd:YAG 1064nm multiplex laser system and electrosurgery.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Able to give informed consent themselves
* Willing to return for follow up visit
* 0.5 - 3 millimeter Vessel size
* 5 Non-contiguous nasal vascular lesions

Exclusion Criteria:

* Mentally handicapped
* Unable to understand written and oral English
* Incarceration
* Under 18 years of age
* Unwilling to return for follow up
* Pregnant Women
* Vessels less than 0.5 millimeter caliber
* Less than 5 non-contiguous vessels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Reduction of Area of Nasal Telangiectasias by Laser Therapy Vs Electrosurgery | 3 months
  The study will measure the changes in length and width (area) of nasal telangiectasias before and after treatment with the following: no treatment (control site), alexandrite laser, pulsed dye laser, combination pulsed dye laser and Nd:YAG 1064nm multiplex laser system and electrosurgery.

SECONDARY OUTCOMES:
Evaluation of Cosmetic Improvement | 3 months
  Percent perceived improvement for nasal vessels by the patient via questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, M.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California-Davis, Department of Dermatology, Sacramento, California, United States

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical